CLINICAL TRIAL: NCT03139149
Title: Comparison of Early Operative Treatment (12 h) and 48 h Conservative Treatment in Acute Small Bowel Obstruction
Brief Title: Comparison of Early Operative Treatment and 48 h Conservative Treatment in Small Bowel Obstruction
Acronym: COTACSO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Alexander E. Tyagunov, MD. Prof, Pirogov Russian National Research Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14121729
Record Dates: First submitted 2017-03-30; First posted 2017-05-03 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Small Bowel Obstruction; Small Bowel Adhesion; Strangulation of Ileum
Keywords: conservative treatment; laparoscopic adhesiolysis; strangulation
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early surgery (Active Comparator): After exclusion of indications for an emergency operation, conservative treatment is performed up to 12 hours from the moment of admission. Each patient receive blood test, blood lactate investigation, blood biochemistry, X-ray of the abdomen, ultrasound and CT on the admission. Each patient receive water-soluble contrast in 3 h after admission. In case of of clinical and radiologic signs of obstruction in 12 h after admission, surgery is performed. On the first stage of surgical treatment laparoscopic adhesiolysis is performed. If it is impossible to eliminate the cause of obstruction by laparoscopic technique laparotomy is performed.
  Interventions: Procedure: Adhesiolysis; Radiation: X-ray diagnostics; Radiation: Computer tomography; Procedure: Ultrasound; Other: General and biochemical blood test
- Late surgery (Active Comparator): After exclusion of indications for an emergency operation, conservative treatment is performed up to 48 hours from the moment of admission. Each patient receive blood test, blood lactate investigation, blood biochemistry, X-ray of the abdomen, ultrasound and CT on the admission. Each patient receive water-soluble contrast 3 h after admission. In case of present of obstruction and absence of contrast in colon in 36 h after intake (48 h after admission) a surgery is perform. On the first stage of surgical treatment laparoscopic adhesiolysis is performed. If it is impossible to eliminate the cause of obstruction by laparoscopic technique laparotomy is performed.
  Interventions: Procedure: Adhesiolysis; Radiation: X-ray diagnostics; Radiation: Computer tomography; Procedure: Ultrasound; Other: General and biochemical blood test

INTERVENTIONS:
Procedure: Adhesiolysis — Method of video laparoscopic operation:
  * Open access in the left upper quadrant of the anterior abdominal wall,
  * Installation of trocars, depending on the prevalence of the adhesion process
  * Assessment of the peritoneal adhesion index
  * Detection of the asleep gut
  * Detection of obstacle area
  * Removing the obstacle without trying to completely eliminate the adhesion process in the abdominal cavity
  If there is no possibility to eliminate the cause of intestinal obstruction laparoscopically laparotomy is performed.
Radiation: X-ray diagnostics — X-ray of the thoracic (1) and abdomen (2-5 times) with water soluble contrast.
Radiation: Computer tomography — Computer tomography of abdomen with iv contrast
Procedure: Ultrasound — Ultrasound of the abdomen (2 times)
Other: General and biochemical blood test — General blood test and biochemical blood test 2 times a day

SUMMARY:
This study will compare the results of early surgery after 12 h conservative treatment and 48 h conservative treatment of adhesive small bowel obstruction.

DETAILED DESCRIPTION:
At the admission patients undergo abdomen x-ray, general and biochemical blood test and computer tomography (CT). After exclusion of indications for an emergency operation, patients are given a water-soluble contrast. Conservative treatment is carring out to 12 hours from admission. All patients with resolution of small bowel obstruction in 12 hours will be excluded from the research. Criteria for obstruction release of conservative treatment 1. No pain 2. Appearance of gas in the colon 3. Decrease of bloating 4. Contrast in the colon. After that, if obstruction is not resolved, randomization is performed. First group undergo surgery. Second group undergo conservative treatment with water-soluble contrast evaluation until 48 hours. In the second group surgery is performed if the conservative treatment is not effective. The results of early and late surgery and the results of conservative treatment in groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

Patients with adhesive small bowel obstruction

Exclusion Criteria:

Early postoperative small bowel obstruction Irreducible hernia Strangulation or peritonitis symptoms Impairment of consciousness Unstable hemodynamics

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-10-11 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantity of patients with obstruction release after conservative treatment | in the 2nd group - 48 hours
  No of patients with success of conservative treatment

SECONDARY OUTCOMES:
Readmission rate in conservative treatment and surgery | 12 months
  12 months readmission rate
30 days mortality | 30 days
  Number of patients who has dead in 30 days after admission
Complications rate | 30 days
  Number of complications rate in groups
Quantity of bowel resection | 156 hours
  Number of patients who undergo bowel resection in groups

CONTACTS AND LOCATIONS:
Locations (1):
- Moscow Clinical Hospital 1, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes